CLINICAL TRIAL: NCT00593333
Title: Intramedullary Nailing of the Femur: A Comparison of the Trochanteric and Piriformis Starting Portals
Brief Title: Intramedullary Nailing of the Femur:Trochanteric vs Piriformis Starting Portals
Acronym: TROCHNAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Theiss, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F030211012
Record Dates: First submitted 2007-12-20; First posted 2008-01-15 (Estimated); Results first posted 2013-11-11 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Femur Fracture
Keywords: Femur Fracture; Intramedullary Nailing; Trochanteric Nailing; Piriformis Starting Portal; Trochanteric Insertion Portal
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, A (Active Comparator): Standard femoral intramedullary nail that utilizes a piriformis fossa portal in the treatment of fractures of the subtrochanteric and diaphyseal shaft regions of the femur.
  Interventions: Device: Antegrade Intramedullary Nail
- 2, B (Experimental): Trigen Trochanteric Femoral Nail (Smith & Nephew, Memphis)using a trochanteric insertion portal in the treatment of fractures of the subtrochanteric and diaphyseal shaft regions of the femur
  Interventions: Device: Trigen Trochanteric Femoral Nail

INTERVENTIONS:
Device: Antegrade Intramedullary Nail — Use of an antegrade intramedullary nail implanted through the Piriformis fossa of the femur. The use of these nails has yielded a union rate of 97 - 99%, and has clearly become the most commonly utilized implant for femur fractures.
  Arms: 1, A
Device: Trigen Trochanteric Femoral Nail — Antegrade intramedullary nails developed with a proximal lateral bend that allows implantation through the greater trochanter rather than the piriformis fossa. This start portal is remarkably easier to locate and may be associated with decreased risk of abductor muscle weakness and pain.
  Other Names: Trigen Trochanteric Femoral Nail, Smith & Nephew, Inc.
  Arms: 2, B

SUMMARY:
This project is designed to determine whether or not the trochanteric insertion portal will show any difference when compared with the piriformis fossa portal in terms of pain and strength of the hip abductor muscles, while allowing faster surgical fixation of the femur fracture.

DETAILED DESCRIPTION:
This project is designed as a prospective, randomized, comparative study between the Trigen Trochanteric Femoral Nail (Smith & Nephew, Memphis) and a standard femoral intramedullary nail that utilizes a piriformis fossa portal in the treatment of fractures of the subtrochanteric and diaphyseal shaft regions of the femur. The hypothesis is that the trochanteric insertion portal will have no difference when compared with the piriformis fossa portal in terms of pain and strength of the hip abductor muscles, while allowing faster surgical fixation of the femur fracture.

Any patient who has sustained a fracture of the femur, is at least 19 years of age, and meets the study's inclusion and exclusion criteria will be asked to participate in the study. After informed consent has been obtained, the patient will be taken to the Operating Theater for surgical fixation of the femur fracture. No fracture will be entered into the study unless antegrade femoral nailing is the treatment of choice of the attending surgeon.

The outcome variables consist of the intraoperative and postoperative adverse device effects recorded in the medical record and on the study data collection form, intraoperative and postoperative complications recorded in medical record and on the study data collection form, hip functional outcome using the WOMAC score recorded for each patient, SF-36 score recorded for each patient, results of clinical examination at 6 weeks, 3, 6, and 12 months recorded in medical record and on the study data collection form, radiographic examination evaluated by two surgeons for the presence of callus and radiographic healing recorded in the medical record and on the study data collection form. Radiographic healing at 6 weeks, 3, 6, and 12 months recorded in the medical record and on the study data collection form. (The injury severity score for all multiple trauma patients recorded on the study data collection form, and soft tissue score according to Gustillo and Anderson for open injuries and according to Tscherne for all closed injuries recorded on the study data collection form. This data will be taken into account relative to the outcome variables). The effects will be measured by clinical examination, radiographic examination, and subjective patient's outcome survey. Additionally, hip abductor muscle strength will be measured and ability to perform one leg stance and hop will be documented at 6 and 12 months.

Data will be collected and entered into EXCEL spreadsheets with double keying for quality control purposes and managed by the Department of Orthopaedic Surgery at the University of Alabama at Birmingham (UAB). After data entry is complete, the file(s) will be copied to diskette and delivered to the UAB Biostatistics statistician for analysis and report generation. The analysis will involve simple descriptive statistics (means, standard deviations, proportions) to assure balance of the treatment groups with respect to relevant variables. T-test will be used to compare the mean times to callus formation and radiographic healing between groups. Analysis of covariance will be performed if there are variables that require adjustment. Growth curve analysis (survival models) and Cox regression procedures will be used to compare the rates of callus formation and/or healing between the two groups. Assumption of proportional hazards in the model will be verified before attempting Cox regression procedures. P-values will be computed using a Mann-Whitney U test for non-parametric data.

ELIGIBILITY:
Inclusion Criteria:

* Fracture patterns of the proximal or middle thirds of the femur that will allow antegrade insertion of a femoral nail
* Adult patient (19 years and older)

Exclusion Criteria:

* Nonunions of the femur
* Pathologic fractures
* Documented prior femur fractures with surgical stabilization with an antegrade nail
* Patients who are pregnant, mentally disturbed, or prisoners
* Inability to comply with protocol
* Patients or family members who are unable or unwilling to sign study consent
* Any fracture too proximal or too distal to use an interlocking screw

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Volgas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States

REFERENCES:
- [Background] Ricci WM, Schwappach J, Tucker M, Coupe K, Brandt A, Sanders R, Leighton R. Trochanteric versus piriformis entry portal for the treatment of femoral shaft fractures. J Orthop Trauma. 2006 Nov-Dec;20(10):663-7. doi: 10.1097/01.bot.0000248472.53154.14. PMID 17106375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started in June 2003. Primary completion date December 2008. Study completion date December 2008. Patients were recruited at University of Alabama at Birmingham.
Groups:
- Standard Treatment: Piriformis fossa entry portal for the antegrade nailing was used for this group. Received either a TRIGEN antegrade femoral nail manufactured by Smith & Nephew (Memphis, Tennessee) or an Antegrade Femoral Nail manufactured by Synthes (West Chester, Pennsylvania)
- Trigen: Trochanteric entry portal for the antegrade nailing was used for this group. These subjects received a TRigen Trochanteric Angegrade Nail (TAN) manufactured by Smith & Nephew that incorporates a 4 degree valgus bend in the proximal aspect of the nail.
Period: Overall Study
Arm/Group | Standard Treatment | Trigen
Started | 54 | 56
Completed | 44 | 45
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment: Pirformis fossa entry portal for the antegrade nailing was used for this group. Received either a TRIGEN antegrade femoral nail or an Antegrade Femoral Nail.
- Trigen: Trochanteric entry portal for the antegrade nailing was used for this group. These subjects received a TRigen Trochanteric Angegrade Nail (TAN) that incorporates a 4 degree valgus bend in the proximal aspect of the nail.
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Trigen | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 43 | 40 | 83

OUTCOME MEASURES:

1. Primary Outcome: Healed Femur Fracture
Description: Time to clinically healed fracture as measured by weeks.
Time Frame: baseline to healed fracture (weeks)
Measure: Mean (Full Range); unit: Weeks
Arm/Group | Standard Treatment | Trigen
Number analyzed (Participants) | 44 | 45
Weeks | 31.8 [10.3 to 64.3] | 31.4 [6.3 to 108.1]

ADVERSE EVENTS:
Time Frame: Subjects were followed through 12 months after intervention
Groups:
- Group A: Piriformis fossa entry portal for the antegrade nailing was used for this group. Received either a TRIGEN antegrade femoral nail manufactured by Smith & Nephew (Memphis, Tennessee) or an Antegrade Femoral Nail manufactured by Synthes (West Chester, Pennsylvania)
- Group B: Trochanteric entry portal for the antegrade nailing was used for this group. These subjects received a TRigen Trochanteric Angegrade Nail (TAN) manufactured by Smith & Nephew that incorporates a 4 degree valgus bend in the proximal aspect of the nail.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 3/54 | 1/56
Other Adverse Events (participants affected / at risk) | 7/54 | 8/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=54) | Group B (N=56)
Hematoma requiring surgical intervention (Surgical and medical procedures) | 2 (2) | 1 (1)
Implant failure requiring revision (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=54) | Group B (N=56)
Implant failure not requiring surgical intervention (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Healed with malalignment (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes